CLINICAL TRIAL: NCT00089739
Title: Use of Immune Cell Markers, Cytokines, Transcription Factors and Surface CD Markers as Markers of Ocular Inflammatory Activity
Brief Title: Immune Indicators of Uveitis
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040260; 04-EI-0260
Record Dates: First submitted 2004-08-11; First posted 2004-08-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-10-28

CONDITIONS: GITR; GITR Ligand; Uveitis; Immunosuppression; Suppressor of Cytokine Secretion
Keywords: Uveitis; Suppressor of Cytokine Secretion; GITR; Immunosuppression; GITR Ligand; Intraocular Inflammation
MeSH Terms: conditions — Uveitis

SUMMARY:
This study will try to identify markers of immune activity in uveitis patients that correlate with the state of disease activity. Uveitis is a group of inflammatory eye diseases that can cause vision loss. The study will examine whether certain substances in the blood can predict a reactivation of disease before it occurs, and how therapy may influence the activity of these substances. Previous studies have found some possible markers called GITR (glucocorticoid induced TNF related family receptor), SOCS (suppressors of cytokine secretion), and interleukin-15. Markers such as these may help guide physicians in safely tapering medicines in uveitis patients.

Patients 18 years of age and older with sight-threatening uveitis may be eligible for this study. Participants are slowly tapered off their medicines when their disease is stable and there is no evidence of significant inflammation. If the disease remains inactive during tapering, all drug therapy is eventually stopped. Patients have eye examinations about every 1 to 3 months when the disease is quiet and every 2 to 4 weeks during flare-ups. Blood samples are drawn 2 to 3 times a year. In addition, patients may have the following procedures if needed:

* Eye photography: Eye drops are given to enlarge the pupils for a thorough eye examination, and a special camera is used to take photographs.
* Fluorescein angiography: This test checks for abnormalities of eye blood vessels. A yellow dye is injected into an arm vein and travels to the blood vessels in the eyes. Pictures of the retina are taken with a special camera that flashes a blue light into the eye. The pictures show if any dye has leaked from the vessels into the retina, indicating possible abnormalities.

DETAILED DESCRIPTION:
Indicators of disease activity in supposed autoimmune conditions are actively being sought. We have already described the increased expression of GITR-glucocorticoid induced TNF-related family receptor during active disease and a decrease in its expression when disease activity diminishes. We have preliminary observations in uveitis patients to suggest that suppressors of cytokine activity (SOCS) 1, 3, and 5 may also be active during either a Th1 or Th2 mediated disease. We wish to see if there is a correlation between these markers and whether they can serve as an indicator of impending activation of disease before actual clinical disease, and how therapy may alter their expression. Patients with uveitis will receive standard evaluation and treatment for inflammatory uveitis under this protocol Blood will be drawn when specific clinical criteria are reached for correlation of potential markers with disease activity.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with bilateral sight threatening uveitis requiring systemic immunotherapy who are 18 years and older are eligible. Disease can be active or quiescent, but subjects must be on a minimum prescribed therapy upon enrollment of a dose averaging at least 20 mg/day (or greater than or equal to 0.25 mg/kg/day) of systemic prednisone or a more intensive immunosuppression regimen. More intensive regimens may include from one to three anti-inflammatory treatments for uveitis that include any one of the following (or related) compounds: corticosteroids (including systemic or periorbital administration), topical corticosteroids (when used in combination with other agents), cyclophosphamide, cyclosporine, azathioprine, chlorambucil, tacrolimus, leflunomide, mycophenolate mofetil, or methotrexate.
* Patients who have non-infectious intermediate, posterior, or panuveitis of at least 3 months duration. Included conditions may include but are not limited to intermediate uveitis of the pars planitis subtype, sarcoidosis, the Vogt-Koyanagi-Harada (VKH) syndrome, birdshot retinochoroidopathy, retinal vasculitis and sympathetic ophthalmia.
* Patients who are 18 years of age or older.

EXCLUSION CRITERIA:

Subjects will not be able to enroll if they:

* Are unwilling or unable to give blood at the designated times in the protocol.
* Have another disease or condition affecting vision that will interfere with obtaining study data
* Are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-08-09; Study Completion 2008-10-28

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Li Z, Mahesh SP, Kim BJ, Buggage RR, Nussenblatt RB. Expression of glucocorticoid induced TNF receptor family related protein (GITR) on peripheral T cells from normal human donors and patients with non-infectious uveitis. J Autoimmun. 2003 Aug;21(1):83-92. doi: 10.1016/s0896-8411(03)00085-4. PMID 12892739